CLINICAL TRIAL: NCT02194231
Title: ATREUS Trial - A Phase II Study on the Activity of Trabectedin of Pretreated Epithelioid or Biphasic / Sarcomatoid Malignant Pleural Mesothelioma(MPM)
Brief Title: ATREUS - Phase II Study on the Activity of Trabectedin in Patients With Malignant Pleural Mesothelioma (MPM)
Acronym: ATREUS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mario Negri Institute for Pharmacological Research (Other)
Collaborators: PharmaMar (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRFMN-MPM-6077; 2011-006330-16 (EudraCT Number)
Record Dates: First submitted 2014-07-16; First posted 2014-07-18 (Estimated); Last update posted 2020-01-23 (Actual); Status verified 2020-01

CONDITIONS: Malignant Pleural Mesothelioma
Keywords: Mesothelioma; MPM; Trabectedin
MeSH Terms: conditions — Mesothelioma, Malignant; Mesothelioma | interventions — Trabectedin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Trabectedin (Experimental): Patients will receive trabectedin treatment
  Interventions: Drug: Trabectedin

INTERVENTIONS:
Drug: Trabectedin — Patients will receive 1.1 mg/m2 intravenous trabectedin infusion in 5% glucose via central venous catheter over 3 hours every 21 days. Trabectedin infusion will be preceded by 20 mg of intravenous dexamethasone
  Other Names: Yondelis

SUMMARY:
The purpose of this study is to determine whether trabectedin is effective in the treatment of malignant pleural mesothelioma (MPM).

DETAILED DESCRIPTION:
There are no approved agents for second-line treatment of MPM in patients who failed first line pemetrexed plus platinum derivatives regimens. Chemotherapy options are limited and include gemcitabine, vinorelbine and other antifolate compounds. The role of second-line chemotherapy is therefore not yet established and second-line patient population is considered suitable for phase II studies with investigational agents.

Trabectedin is an originally natural marine product, now obtained by a semisynthetic process, that induces a delay in S phase progression and a blockade in G2 phase of the cell cycle by a mode of action that seems different from that of other DNA-damaging agents (see citations). Although the exact mechanism of action of trabectedin has not been fully elucidated yet, it appears to be unique compared to other anticancer agents (see citations). Trabectedin binds to N2 of guanines in the minor groove of DNA, causing a bending of the minor groove towards the major groove.

In the randomised clinical trials in metastatic leiomyosarcoma or liposarcoma and in recurrent platinum-sensitive ovarian cancer, trabectedin is infused at 1.5 mg/m2 as a 24-hour infusion or 1.3 mg/m2 as a 3 hour infusion every 3 weeks (see citations). Balancing efficacy with safety the short infusion is preferable in clinical practice.

In soft tissue sarcoma the response rate did not exceed 10%, however, trabectedin has been shown to provide disease control, with progression arrest rates exceeding 50% and progression-free survival rates exceeding 20% at 6 months. In pre-treated ovarian cancer the objective response rate was 30% with a median time to disease progression of 5.7 months.

Trabectedin has not been extensively employed in MPM, however in phase I studies, some objective response in heavily pre-treated mesothelioma patients was seen.

The present study is aimed at evaluating the activity of trabectedin in MPM patients not candidate for radical surgery. This option is of particular interest due to lack of valid therapeutic options.

Translational studies will be performed to identify factors predictive of the activity of trabectedin in MPM.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically proven unresectable MPM. In order to make a reproducible diagnosis, in particular regarding biphasic MPM, histology must derive from transthoracic biopsies (at least 3 representative samples) or from videothoracoscopy (at least 5 representative samples)
2. Age >18 years
3. Performance status 0-1 (ECOG)
4. Measurable disease (CT-PET) according to RECIST criteria modified for malignant pleural mesothelioma
5. Not more than one previous chemotherapy course (consisting of pemetrexed plus platinum derivative), excluded adjuvant therapy if PFS < 12 months
6. A minimum of 3 weeks since previous tumour directed therapy
7. Recovery from toxic effects of previous therapies to NCI CTC AE Grade 0-1
8. Patients who have received palliative radiation are eligible if <30% of bone marrow was irradiated and normal haematological function was completely regained
9. Haematologic variables: haemoglobin ≥ 9 g/dL, Absolute neutrophil count (ANC) ≥ 1,500/μL and Platelet count ≥ 100,000/μL
10. Serum creatinine ≤1.5 mg/dL or creatinine clearance ≥ 30 mL/min
11. Creatinine phosphokinase (CPK) ≤ 2.5 ULN
12. Hepatic function variables: Total bilirubin ≤ ULN, Total alkaline phosphatase ≤ 2.5 ULN or if > 2.5 ULN alkaline phosphatase liver fraction or GGT or 5' nucleotidase must be determined and ≤ ULN, AST (serum aspartate transaminase [SGOT]) and ALT (serum alaninetransaminase [SGPT]) must be ≤ 2.5 x ULN, Albumin ≥ 25 g/L
13. Signed informed consent
14. Adequate contraceptive methods for male patients whose partner is of childbearing age/potential, during the study and for three months after the end of treatment

Exclusion Criteria:

1. - Radiotherapy with curative intent to thoracic wall (concomitant with or prior to chemotherapy)
2. - Uncompensated diabetes mellitus or other condition absolutely contra-indicating dexamethasone (used as pre-medication)
3. - Patients enrolled in other study with experimental drugs
4. - Women of childbearing age/potential
5. - Prior exposure to trabectedin
6. - History of other malignancies (except basal cell carcinoma or cervical carcinoma in situ, adequately treated), unless in remission from 5 years or more and judged of negligible potential of relapse
7. - Active viral hepatitis or chronic liver disease
8. - Unstable cardiac condition, including congestive heart failure or angina pectoris, myocardial infarction within one year before enrolment, uncontrolled arterial hypertension or arrhythmias
9. - Active major infection
10. - Other serious concomitant illness
11. - Brain / leptomeningeal involvement

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 145 (Actual)
Dates: Start 2013-07; Primary Completion 2019-12-12 (Actual); Study Completion 2019-12-12 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival - PFS12w | 12 weeks
  Proportion of patients free from progression or death at the second CT scan assessment performed at 12 weeks (Progression Free Survival - PFS12w) from the date of treatment start

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | 24 months
  PFS will be evaluated by CT scans every 6 weeks from the date of first treatment until week 12 and subsequently every 8-9 weeks
Overall survival (OS) | 24 months
Objective response rate | 24 months
  Responses will be assessed according to Modified RECIST criteria for Malignant Pleural Mesothelioma
Trabectedin tolerability and safety | 24 months
  Safety will be evaluated based on reported AEs, clinical laboratory assessments, vital signs and physical examinations. Adverse events will be encoded using the Medical Dictionary for Regulatory Activities (MedDRA) and graded using NCI-CTCAE ver 4
Pain Intensity (PI) | 24 months
  Pain intensity will be evaluated by using an 11 points Numerical Rating Scale (NRS), where 0 indicates no pain and 10 indicates the worst pain one can imagine. Patients will be requested to evaluate the PI related to the 24 hours preceding the visit and indicating the score for the average, worst and least PI
Pain type and characteristics | 24 months
  With special reference to the presence of neuropathic pain, evaluation shall be carried out using the DN4 questionnaire. The global score on this 10 item instrument allows to diagnose the presence of neuropathic pain (total score ≥4)
Antalgic treatments | 24 months
  Evaluation of type and dosage of any pain medication administered to the patient at the moment of the study visit
microRNA (miRs) profile | 24 months
  miRs profile evaluation will be performed with the aim of characterising the tumour biological features associated to the different response patterns. Since recent published studies suggests that trabectedin modulates the expression of some miRs in cancer cells exposed to the drug and, also, the resistance to anticancer drugs seems to be well correlated to the expression of some specific miRs, the evaluation of miRs expression may become a powerful prognostic and predictive marker.
  miRNA landscape in both plasma and tumour tissues will be profiled using commercially available oligo arrays platforms.
High Mobility Group B1 (HMGB1) protein assessment | 24 months
  Recent data indicate that the high mobility group B1 (HMGB1) is implicated in the transformation of meshothelial cells and is strongly secreted in sera of patients with mesothelioma. These findings provide the rationale for considering HMGB1 as a potential useful marker to monitor therapeutic effectiveness in patients with mesothelioma.
  HMGB1 will be determined in plasma of patients at the same time points previously indicated for the assessment of miR profiles by using an ELISA essay
Blood Macrophages analysis | 24 months
  We propose to analyse the effects of trabectedin on the number of circulating monocytes and the plasma levels of selected biological mediators. A decrease in the number of circulating monocytes could be a surrogate marker of a biological effect of trabectedin on the precursor cells of tumour macrophages.
  We propose to collect the number of circulating monocytes during the first 3 treatment cycles, immediately before and 7 days after trabectedin administration

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Bidoli, MD, Principal Investigator — Azienda Ospedaliera San Gerardo di Monza; Valter Torri, MD, Study Chair — Istituto Di Ricerche Farmacologiche Mario Negri
Locations (8):
- Italy (8):
  - Azienda ospedaliera ss. Antonio e Biagio e Cesare Arrigo, Alessandria, AL
  - Cliniche Humanitas Gavazzeni, Bergamo, BG
  - Azienda Ospedaliera Universitaria Policlinico Sant'Orsola Malpighi, Bologna, Bo
  - P.O. Spedalli Civili, Brescia, BS
  - Azienda Ospedaliera S. Gerardo di Monza, Monza, MB
  - Istituto Clinico Humanitas, Rozzano, MI
  - Istituto Oncologico Veneto - IOV, Padua, PD
  - Azienda Ospedaliro-Universitaria di Parma, Parma

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Pommier Y, Kohlhagen G, Bailly C, Waring M, Mazumder A, Kohn KW. DNA sequence- and structure-selective alkylation of guanine N2 in the DNA minor groove by ecteinascidin 743, a potent antitumor compound from the Caribbean tunicate Ecteinascidia turbinata. Biochemistry. 1996 Oct 15;35(41):13303-9. doi: 10.1021/bi960306b. PMID 8873596
- [Result] Bonfanti M, La Valle E, Fernandez Sousa Faro JM, Faircloth G, Caretti G, Mantovani R, D'Incalci M. Effect of ecteinascidin-743 on the interaction between DNA binding proteins and DNA. Anticancer Drug Des. 1999 Jun;14(3):179-86. PMID 10500494
- [Result] Erba E, Bergamaschi D, Bassano L, Damia G, Ronzoni S, Faircloth GT, D'Incalci M. Ecteinascidin-743 (ET-743), a natural marine compound, with a unique mechanism of action. Eur J Cancer. 2001 Jan;37(1):97-105. doi: 10.1016/s0959-8049(00)00357-9. PMID 11165136
- [Result] Demetri GD, Chawla SP, von Mehren M, Ritch P, Baker LH, Blay JY, Hande KR, Keohan ML, Samuels BL, Schuetze S, Lebedinsky C, Elsayed YA, Izquierdo MA, Gomez J, Park YC, Le Cesne A. Efficacy and safety of trabectedin in patients with advanced or metastatic liposarcoma or leiomyosarcoma after failure of prior anthracyclines and ifosfamide: results of a randomized phase II study of two different schedules. J Clin Oncol. 2009 Sep 1;27(25):4188-96. doi: 10.1200/JCO.2008.21.0088. Epub 2009 Aug 3. PMID 19652065
- [Result] Del Campo JM, Roszak A, Bidzinski M, Ciuleanu TE, Hogberg T, Wojtukiewicz MZ, Poveda A, Boman K, Westermann AM, Lebedinsky C; Yondelis Ovarian Cancer Group. Phase II randomized study of trabectedin given as two different every 3 weeks dose schedules (1.5 mg/m2 24 h or 1.3 mg/m2 3 h) to patients with relapsed, platinum-sensitive, advanced ovarian cancer. Ann Oncol. 2009 Nov;20(11):1794-802. doi: 10.1093/annonc/mdp198. Epub 2009 Jun 25. PMID 19556318
- [Result] D'Incalci M, Galmarini CM. A review of trabectedin (ET-743): a unique mechanism of action. Mol Cancer Ther. 2010 Aug;9(8):2157-63. doi: 10.1158/1535-7163.MCT-10-0263. Epub 2010 Jul 20. PMID 20647340